CLINICAL TRIAL: NCT04466215
Title: Medication Development for Protracted Abstinence in Alcoholism: CORT118335 Versus Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NIAAAMAS006420; U01AA025476 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol-Related Disorders
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders | interventions — CORT118335; Sugars

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Double-Blind, Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Miricorilant (Active Comparator): 900 mg (6 x 150 mg) tablets daily taken orally for two weeks
  Interventions: Drug: Miricorilant
- Placebo (Placebo Comparator): Six placebo tablets taken orally for two weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Miricorilant — 900 mg (6 x 150 mg) tablets taken orally once daily for two weeks
  Other Names: CORT118335
  Arms: Miricorilant
Drug: Placebo oral tablet — Six placebo tablets taken orally once daily for two weeks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The hypotheses under test are that subjects with alcohol use disorder (AUD) of moderate or greater severity treated with CORT118335 will report decreased craving for alcohol following alcohol exposure in the laboratory and report significantly less drinking under naturalistic conditions, than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-75 years of age.
* Meets DSM-5 criteria for current alcohol use disorder of moderate or greater severity (AUD-MS).
* Subjects will not be seeking treatment because the medication studies are not treatment trials, and to avoid exposing treatment-seekers to alcohol cues.
* Subjects must be abstinent a minimum of 3 days (but not more than 7 days) prior to the human lab session.
* In acceptable health in the judgment of the study physician, based on interview, medical history, physical exam, ECG, routine urine and blood chemistry.
* Subjects with a history of depression, who have been on a stable dose of anti-depressant medication for at least 3 months, and do not meet current DSM-5 criteria for depression or anxiety.
* All subjects must agree to use double barrier birth control for the study duration and one month thereafter i.e., males must use condoms and females must use spermicide and/or a non hormonal barrier method, and their opposite sex partner must likewise use an effective non hormonal form of contraception.
* Able to provide informed consent and understand questionnaires and study procedures in English.
* Willing to comply with the provisions of the protocol and take daily oral medication

Exclusion Criteria:

* Medical conditions that could be aggravated by glucocorticoid and/or mineralocorticoid antagonism.
* Clinically significant findings on physical exam, ECG, urine or blood tests that may increase risk.
* CYP2C19 inhibitors
* Substrates metabolized primarily by CYP3A, CYP2C9, and CYP2C8 with narrow therapeutic index
* BCRP and UGT1A1 substrates
* Meets DSM-5 criteria for a current major psychiatric disorder, including mood, anxiety or substance use disorders, other than alcohol, nicotine, or mild cannabis use disorders.
* Pregnant or lactating.
* Treatment within the month prior to screening with (1) an investigational drug, (2) drugs which may negatively interact with study medications, or (3) drugs that may influence study outcomes (e.g., disulfiram [Antabuse], naltrexone [ReVia], acamprosate [Campral], or anticonvulsants.
* Chronic systemic steroid use
* Using drugs that are strong inhibitors and inducers of CYP2C9.
* No fixed domicile and/or no availability by home or mobile telephone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute Pearson Center for Alcoholism and Addiction Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, CA from 04/15/2021-05/25/2022. Seventy-seven non-treatment seeking, paid volunteers signed informed consent, Fifty subjects were enrolled, and Fifty subjects completed the study.
Pre-assignment Details: Twenty-seven subjects were excluded from study participation, twenty-five did not meet admission criteria and two declined to participate.
Groups:
- CORT118335: 900 mg (6 x 150 mg) tablets daily taken orally for two weeks
  CORT118335: 900 mg (6 x 150 mg) tablets taken orally once daily for two weeks
Period: Overall Study
Arm/Group | CORT118335 | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CORT118335 | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.04 (12.9) | 43.56 (15.0) | 42.3 (28.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 18 | 21 | 39
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
DSM-V symptom count [Mean (Standard Deviation); unit: Symptom count] — Symptom count from the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria for Alcohol Use Disorder (AUD)
  Symptom count | 6.56 (1.9) | 6.56 (1.5) | 6.56 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Craving to Drink
Description: Total Visual Analog Scale (VAS) scores of craving severity in response to in vivo alcohol cues. Higher scores indicate greater craving severity with a minimum score of 0 and a maximum score of 80.
Time Frame: 1 hour on the last day of dosing (Day 14)
Population: All subjects who completed cue exposure testing in the laboratory were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CORT118335 | Placebo
Number analyzed (Participants) | 25 | 24
score on a scale | 31.1 [23.8 to 38.5] | 33.2 [23.3 to 43.0]
Statistical Analysis 1: Comparison: CORT118335 vs Placebo; Mixed effect model with directional hypothesis that drug reduces strength of craving (VAS). Principle predictor was drug plasma concentration. Arms were combined for this analysis; Test type: Superiority; p = .065, Mixed Models Analysis — One-tail test of directional hypothesis; Slope = -0.063, Standard Error of Mean .04

2. Secondary Outcome: Drinking
Description: Number of standard drinks per day using the Timeline Followback Interview (TLFB). Total number of alcoholic drinks consumed per day with a minimum value of 0 and an undetermined maximum value.
  Treatment effects on drinking were assessed during the 11 days of ad libitum drinking and did not include the final three days of mandatory abstinence prior to cue reactivity session.
Time Frame: 11 days (Treatment effects on drinking were assessed during the 11 days of ad libitum drinking)
Population: All subjects with post baseline drinking data were included.
Measure: Mean (Standard Error); unit: Average drinks per day
Arm/Group | CORT118335 | Placebo
Number analyzed (Participants) | 25 | 25
Average drinks per day | 3.7 (.41) | 3.7 (.29)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all study visits, for an average duration of 4 weeks (2 weeks on drug, and 2 weeks post treatment).
Description: Adverse events, both serious and other, were documented at all study visits by the Medical Assistant on the adverse events case report form.
Arm/Group | CORT118335 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 9/25 | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CORT118335 (N=25) | Placebo (N=25)
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Fatigue (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 2
Feeling less euphoric (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04466215/Prot_003.pdf
  • Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT04466215/SAP_004.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04466215/ICF_005.pdf